CLINICAL TRIAL: NCT02589600
Title: ZEST II for Osteoporotic Fracture Prevention
Brief Title: Zoledronic Acid for Osteoporotic Fracture Prevention (ZEST II)
Acronym: ZEST II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Susan L. Greenspan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Susan L. Greenspan, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19040149 (ZEST II); 1R01AG050302-01A1 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Osteoporotic Fractures; Osteoporosis, Postmenopausal
Keywords: Bone loss; Frail Geriatric Women; Nursing Home Patients; Long-term Care Patients; Osteoporosis; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Osteoporosis | interventions — Zoledronic Acid; Vitamin D; Calcium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Medication Group (Experimental): Annual dose: intravenous zoledronic acid (Reclast) 5.0 mg; vitamin D (800 IU/daily) and calcium (approximately 1200 mg/daily, dietary + supplements)
  Interventions: Drug: Zoledronic acid; Dietary Supplement: vitamin D; Dietary Supplement: calcium
- Placebo Group (Placebo Comparator): Annual dose: intravenous saline; vitamin D (800 IU/daily and calcium (approximately 1200 mg/daily, dietary + supplements)
  Interventions: Dietary Supplement: vitamin D; Dietary Supplement: calcium; Other: Saline

INTERVENTIONS:
Drug: Zoledronic acid — Annual intravenous 5.0 mg
  Other Names: Reclast
  Arms: Active Medication Group
Dietary Supplement: vitamin D — 800 IU daily
Dietary Supplement: calcium — approximately 1200 mg (dietary and supplement)
Other: Saline — Annual intravenous saline placebo
  Arms: Placebo Group

SUMMARY:
The goal of this study is to perform the first fracture reduction clinical trial with a potent antiresorptive agent (intravenous zoledronic acid) in the most vulnerable long-term care population.

DETAILED DESCRIPTION:
Although close to 85% of frail women in long-term care (LTC) facilities have osteoporosis and the risk of osteoporotic fractures is nearly 10 times that of community dwelling elderly, few are treated and studies are scarce. It is postulated that in frail, LTC women an annual infusion of zoledronic acid, an antiresorptive therapy for osteoporosis, will:

1. be effective demonstrated by fracture reduction;
2. be safe.

To address these hypotheses, up to 1000 female LTC residents age 65 and older will be screened in order to enroll 310 eligible for randomization in a 3 year, randomized, double-blind, calcium and vitamin D controlled trial with the antiresorptive agent zoledronic acid. Use of an intravenous, once yearly agent avoids concerns of oral bisphosphonate side effects, poor absorption and burden on staff. Participants will reside in the long-term care settings associated with the Division of Geriatric Medicine, University of Pittsburgh and will include women with multiple comorbid conditions, functional and cognitive impairment, and limited mobility.

ELIGIBILITY:
Inclusion Criteria:

* women age ≥65 years including those using assistive devices to maximize generalizability if they:

  1. Reside in long-term care (LTC);
  2. Have:

     * osteoporosis by axial bone density (spine, hip or forearm bone mineral density (BMD) T-score ≤ -2.5 SD); or
     * a previous adult fragility fracture of the spine or hip; or,
     * would be treated based on FRAX National Osteoporosis Foundation (NOF) treatment thresholds of a 10 year risk of ≥ 20% for a major osteoporotic fracture or ≥ 3% for hip fracture using femoral neck BMD.

Exclusion Criteria:

* Men because osteoporosis is less common in men and our initial ZEST 1 study only included women.
* Institutionalized women with subacute illnesses surviving or discharged in < 3 years.
* Women currently on bisphosphonate, denosumab, or teriparatide therapy or who have been on a bisphosphonate for greater than 1 year during the previous 2 years because bisphosphonates are long acting.
* Patients with a calculated creatinine clearance < 35 ml/min or who have a contraindication for bisphosphonates (allergy, hypocalcemia).

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 310 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Osteoporosis Prevention & Treatment Center, New Kensington, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will occur during the first 2 years of the grant cycle and take place in the determined long term care facilities.
Pre-assignment Details: 310 subjects were consented, randomized and received the study drug.
Period: Overall Study
Arm/Group | Active Medication Group | Placebo Group
Started | 154 | 156
Completed | 101 | 102
Not Completed | 53 | 54

BASELINE CHARACTERISTICS:
Population: Same as participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Medication Group | Placebo Group | Total
Number analyzed (Participants) | 154 | 156 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 154 | 156 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.3 (7.9) | 79.9 (7.7) | 80.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 156 | 310
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 151 | 155 | 306
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 142 | 146 | 288
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 154 | 156 | 310

OUTCOME MEASURES:

1. Primary Outcome: Non-traumatic Incidental Fractures (Vertebral and Nonvertebral [Identified by X-ray, CT, MRI, VFA Imaging] Per Person-year)
Description: Number of fractures divided by number of person-years. Effectiveness of fracture reduction will be demonstrated by total non-traumatic incidental fractures (vertebral and nonvertebral [identified by x-ray, CT, MRI, VFA imaging) except those viewed as severe trauma (fall from a height higher than a stool or chair or severe trauma other than a fall), cancer-related or fractures of the toes, finger or facial bones.
Time Frame: 3 years
Population: Women age 65 years and older
Measure: Number; unit: Fractures per person-year
Arm/Group | Active Medication Group | Placebo Group
Number analyzed (Participants) | 154 | 156
Fractures per person-year | 1.06093 | 1.01563
Statistical Analysis 1: Comparison: Active Medication Group vs Placebo Group; Test type: Superiority; p = 0.7251, Negative binomial regression; Incident Rate Ratio = 1.05, 95% CI 2-sided [.90 to 1.22] — Placebo group is the reference group; Negative binomial regression implemented in the SAS®️ GENMOD procedure with fracture outcome as the dependent variable; duration of follow-up as an offset to account for each participant's exposure; treatment arm as the main independent factor of interest

ADVERSE EVENTS:
Time Frame: Up to three years.
Arm/Group | Active Medication Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 13/154 | 19/156
Serious Adverse Events (participants affected / at risk) | 73/154 | 80/156
Other Adverse Events (participants affected / at risk) | 131/154 | 130/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Medication Group (N=154) | Placebo Group (N=156)
Anemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 5
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 5
Chest pain (Cardiac disorders) | 8 | 7
Edema peripheral (Cardiac disorders) | 0 | 1
Fluid overload (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0
Hypoglycemia (Endocrine disorders) | 2 | 0
Blurred vision (Eye disorders) | 0 | 1
Microvascular cranial nerve palsy (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal Spasm (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 3
Diarrhea hemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 4
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 5 | 6
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 13 | 19
Gait disturbance (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Weakness (General disorders) | 5 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bacteremia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 3
COVID-19 (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 4 | 4
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 9 | 7
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Hematoma (Injury, poisoning and procedural complications) | 4 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Fractured sacrum (Musculoskeletal and connective tissue disorders) | 0 | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 6 | 4
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Patella Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Pubic rami fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Radius fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Thoracic vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Confusional state (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 3
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Ischemic cerebral infarction (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Normal Pressure Hydrocephalus (Nervous system disorders) | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 6 | 2
Transient ischemic attack (Nervous system disorders) | 4 | 1
Vertigo positional (Nervous system disorders) | 1 | 0
Acute Confusional State (Psychiatric disorders) | 1 | 4
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 4 | 8
Adenoviral upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lobar Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cellulitis (Skin and subcutaneous tissue disorders) | 3 | 3
Aortic Valve replacement (Surgical and medical procedures) | 0 | 1
Colectomy (Surgical and medical procedures) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Hernia hiatus repair (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 4 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 3
Mastectomy (Surgical and medical procedures) | 2 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 0
Oesophagogastric fundoplasty (Surgical and medical procedures) | 0 | 1
Open reduction of fracture (Surgical and medical procedures) | 0 | 1
Rectal Prolapse Repair (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 3
Spinal laminectomy (Surgical and medical procedures) | 2 | 1
Thromboembolectomy (Surgical and medical procedures) | 1 | 0
Vaginal fistula repair (Surgical and medical procedures) | 0 | 1
skin graft (Surgical and medical procedures) | 0 | 2
Aortic Dissection (Vascular disorders) | 0 | 1
Aortic Stenosis (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
Lymphedemas (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Medication Group (N=154) | Placebo Group (N=156)
Chest pain (Cardiac disorders) | 8 | 7
Fall (Injury, poisoning and procedural complications) | 9 | 7
Urinary tract infection (Renal and urinary disorders) | 16 | 17
Atrial fibrillation (Cardiac disorders) | 7 | 8
Diarrhea (Gastrointestinal disorders) | 15 | 18
Nausea (Gastrointestinal disorders) | 22 | 14
Vomiting (Gastrointestinal disorders) | 9 | 3
Fatigue (General disorders) | 15 | 10
Influenza like illness (General disorders) | 22 | 9
Fall (Injury, poisoning and procedural complications) | 59 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 17
Dizziness (Nervous system disorders) | 3 | 13
Headache (Nervous system disorders) | 30 | 18
Cellulitis (Skin and subcutaneous tissue disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02589600/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02589600/SAP_001.pdf
  • Informed Consent Form (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02589600/ICF_002.pdf